CLINICAL TRIAL: NCT01371877
Title: The Role of Vitamin D in Chronic Urticaria and Angioedema Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0271-11-FB
Record Dates: First submitted 2011-06-01; First posted 2011-06-13 (Estimated); Results first posted 2014-12-16 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Urticaria; Angioedema; Hives; Swelling
Keywords: urticaria; angioedema; hive; swelling
MeSH Terms: conditions — Urticaria; Angioedema | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 4000 IU (Experimental): Subjects will be randomized 1:1 to high dose vitamin D defined as 4000 IU per day for 3 months.
  Subjects will be given Vitamin D3 supplementation at 4000 IU daily.
  Interventions: Drug: High Dose Vitamin D3
- Vitamin D3 600 IU (Active Comparator): Subjects will be randomized 1:1 to low dose vitamin D as defined as 600 IU per day for 3 months.
  Subjects will be given Vitamin D3 supplementation at 600 IU daily
  Interventions: Drug: Low Dose Vitamin D3

INTERVENTIONS:
Drug: High Dose Vitamin D3 — Vitamin D 4000 IU per day for 3 months
  Other Names: cholecalciferol
  Arms: Vitamin D3 4000 IU
Drug: Low Dose Vitamin D3 — Vitamin D 600 IU per day
  Other Names: cholecalciferol
  Arms: Vitamin D3 600 IU

SUMMARY:
This clinical study was designed based on our hypothesis that vitamin D plays an important role in chronic urticaria and that high dose supplementation with vitamin D in subjects with chronic urticaria will improve clinical response.

This clinical study will investigate our hypothesis in three Specific Aims:

1. Determine whether high dosing vitamin D supplementation (4000 IU/day) reduces medication usage (primary outcome) and urticaria severity score (secondary outcome) in subjects with chronic urticaria as compared to low dosing (600 IU/day).
2. Determine if high dosing of vitamin D (4000 IU/day) is safe and well-tolerated in subjects with chronic urticaria with or without baseline vitamin D deficiency.
3. Investigate whether there is an association with serum 25-hydroxyvitamin D levels, vitamin D receptor mRNA expression, and chronic urticaria severity.

DETAILED DESCRIPTION:
The purpose of this pilot, 12 week, clinical research study is to determine if supplementation with Vitamin D will improve the clinical outcome in subjects with chronic urticaria and angioedema (CUA). Vitamin D is a key element in the regulation of immune system responses, and vitamin D could play an important role in the treatment of CUA. Recently, we published that there is an important association with CUA and serum 25-hydroxy vitamin D (25OHD). Namely, vitamin D levels in subjects with CUA were significantly lower as compared to subjects with an alternative allergic disorder, allergic rhinitis. There is now one other observational report that supplementation with vitamin D (50,000/wk) in subjects CUA resulted in clinical improvement; however, there was only one treatment arm and optimal serum 25OHD required to obtain benefit was not investigated.

This current study is a double-blinded, prospective, interventional study that seeks to recruit adult subjects with physician-diagnosed CUA and randomize subjects to either the recommended dietary allowance (Vitamin D 600 IU/day) or the recommended upper limit of intake (Vitamin D 4000 IU/day). Subjects will answer a questionnaire to collect information regarding demographics, previous diagnostic tests, medications, and complete an urticaria severity score (USS). Information from the medical record: weight, height, body mass index (BMI), thyroid stimulating hormone (TSH), free thyroxine (T4), thyroid autoantibodies, urticaria autoimmune testing (CD203c results), anti-nuclear antibody (ANA), urinalysis, and allergy skin prick testing, which are part of the CUA evaluation will be obtained. Subjects will have research blood draws for serum 25OHD level, iPTH, calcium, phosphorus, albumin, urine calcium, and vitamin D receptor (VDR) gene expression. All subjects will receive standard-of-care therapy according to the 2009 Third International Consensus Meeting on Urticaria position guidelines. Follow-up visits for medication usage, urticaria severity score, and serum and urine safety monitoring will be at 6 and 12 weeks.

The hypothesis of this study is that high dosing of vitamin D will result in clinical improvement in subjects with CUA. The primary clinical endpoint is medication usage, and the secondary outcomes are urticaria severity score and prednisone rescue use. We will explore if threshold serum 25OHD levels correlate and VDR expression correlate to clinical outcomes, and to determine power analysis to conduct a larger scale study. Finally, the study aims to determine if vitamin D supplementation is safe and well-tolerated in subjects with CUA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included if they have physician-diagnosed chronic urticaria and/or angioedema (CUA). CUA is defined by having urticarial wheals (hives) and/or angioedema (dermal swelling) on a daily or almost daily for more than 6 weeks. Patients with CUA also having signs of dermatographism and/or delayed-pressure urticaria will be included in the study. Subjects with history of intolerance to non-steroidal anti-inflammatory drugs will be included but warned not to take this drug class (acetaminophen will be allowed instead).

Exclusion Criteria:

* Subjects will be excluded if:

  1. They are not capable of answering the questionnaire.
  2. Subjects with a pure physical or allergic urticarias, and/or hereditary and acquired angioedema (C1 esterase inhibitor deficiency). These subjects will be excluded as the etiology of their disease is known.
  3. Pregnant or lactating women. All child-bearing women will be asked (verbally and on the questionnaire) if they are pregnant or lactating. If they answer yes, they will be excluded. As there is no risk or harm to the pregnant or lactating woman, a urine pregnancy test will not be used.
  4. Subjects with any clinically significant abnormality in biochemistry testing, and/or hypercalcemia (calcium > 10.3 mg/dl) or renal insufficiency (GFR< 50 ml/min).
  5. Subjects with a history of primary hyperparathyroidism, renal tubular acidosis, sarcoidosis, granulomatous disease, or malignancy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2013-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill A Poole, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Thorp WA, Goldner W, Meza J, Poole JA. Reduced vitamin D levels in adult subjects with chronic urticaria. J Allergy Clin Immunol. 2010 Aug;126(2):413; author reply 413-4. doi: 10.1016/j.jaci.2010.04.040. No abstract available. PMID 20621341
- [Derived] Rorie A, Goldner WS, Lyden E, Poole JA. Beneficial role for supplemental vitamin D3 treatment in chronic urticaria: a randomized study. Ann Allergy Asthma Immunol. 2014 Apr;112(4):376-82. doi: 10.1016/j.anai.2014.01.010. Epub 2014 Feb 5. PMID 24507460

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Vitamin D: Subjects will be randomized 1:1 to high dose vitamin D defined as 4000 IU per day for 3 months.
  Vitamin D: Vitamin D 4000 IU per day for 3 months
- Low Dose Vitamin D: Subjects will be randomized 1:1 to low dose vitamin D as defined as 600 IU per day for 3 months.
  Vitamin D: Vitamin D 600 IU per day
Period: Overall Study
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D
Started | 21 | 21
Completed | 21 | 17
Not Completed | 0 | 4
Not completed — 3 for unknown reasons and 1 pregnant | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Full Range); unit: years] | 43.9 [19 to 79] | 43.1 [20 to 72] | 43.5 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42
Baseline vitamin D level [Mean (Standard Deviation); unit: ng/mL] | 28.86 (10.1) | 37.2 (15.5) | 33.0 (13.6)

OUTCOME MEASURES:

1. Primary Outcome: Medication Usage
Description: The Unit of Measure is Efficacy. The primary outcome of this study is to determine if vitamin D supplementation reduces the medication usage in subjects with CUA. Thus, for the outcome of reduction in pills, at 12 weeks, subjects whose pill usage decreases by 2 or more pills per day will be classified as improved. Subjects whose pill consumption did not change or increased will be classified as unchanged.
Time Frame: 12 week intervention
Measure: Mean (Standard Deviation); unit: number of pills/day
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D
Number analyzed (Participants) | 21 | 17
number of pills/day
  Baseline medication usage | 2.8 (2.6) | 4.6 (3.2)
  3 month medication usage | 2.0 (2.9) | 4.9 (2.8)

2. Secondary Outcome: Total Urticaria Severity Score at 3 Months
Description: The Unit of Measure is Efficacy. The Total Urticaria Severity Score (USS) ranges from 0 to 93, higher scores = worse symptoms. This secondary outcome of this study is to determine if high dose vitamin D supplementation improves the urticaria severity score (USS). The change in USS will be compared between the groups using the independent sample t-test (assuming the distribution is normal). Logistic regression and multiple linear regression will be used to adjust for possible confounders.
Time Frame: 3 month intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D
Number analyzed (Participants) | 21 | 17
units on a scale
  Baseline Total Urticaria Score | 41.14 (2.36) | 40.1 (3.4)
  1 week Total Urticaria Score | 25.48 (3.34) | 29.24 (3.93)
  3 month Total Urticaria Score | 15.0 (2.9) | 24.1 (2.9)

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Unit of Measure is Safety and Tolerability. The number of participants with adverse events will be compared between the groups using the independent sample t-test (assuming the distribution is normal).
Time Frame: 3 month study trial
Population: No significant adverse events. All subjects in the high vitamin D3 group completed the study; 4 subjects in the low vitamin D3 600 IU/day withdrew from the study (1 for pregnancy and 3 unknown). There was no evidence of hypercalcemia.
Measure: Number; unit: participants
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D
Number analyzed (Participants) | 21 | 21
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected continuously and reported to data safety board every 3 months.
Arm/Group | High Dose Vitamin D | Low Dose Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes